CLINICAL TRIAL: NCT02773654
Title: 1) Mobile Application Utilization for Measurement of Scapular Position 2) 3D Shoulder Motion Measurement Device (The MnMotion System)
Brief Title: Mobile Application Utilization for Measurement of Scapular Position
Acronym: MnMotion
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1604M86268
Record Dates: First submitted 2016-05-10; First posted 2016-05-16 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Shoulder Pain
Keywords: shoulder; motion; measurement; healthy shoulder; shoulder motion
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Asymptomatic subjects: subjects without complaints or history of shoulder pain or obvious movement abnormalities.
  Interventions: Other: Healthy Volunteers
- Symptomatic Volunteers: Symptomatic subjects: subjects with shoulder pain who have active range of motion beyond 120° of elevation.
  Interventions: Other: Symptomatic Volunteers

INTERVENTIONS:
Other: Healthy Volunteers — Scapula static position of subjects with and without shoulder symptoms will be recorded utilizing a mobile phone application placed on their scapula by either the examiner's hands or with a handle, held by the examiner.
  Groups: Healthy Volunteers
Other: Symptomatic Volunteers — Scapula static position of subjects with and without shoulder symptoms will be recorded utilizing a mobile phone application placed on their scapula by either the examiner's hands or with a handle, held by the examiner.
  Groups: Symptomatic Volunteers

SUMMARY:
The purpose of this study is to determine the ability of a mobile clinical application to reliably and accurately track scapular motion in people with asymptomatic and symptomatic shoulders. The ability to accurately and reliably measure shoulder position clinically is an important first step in choosing the best treatment techniques to treat shoulder movement dysfunction. Therefore, the primary objectives of the study are:

1. To determine the inter- and intra-rater reliability of shoulder joint position measurements in symptomatic and asymptomatic subjects, by using a mobile application, with and without use of a handle for a smartphone
2. To determine the validity of the shoulder joint position measurements measurements as described above.

DETAILED DESCRIPTION:
Subjects will be asked to provide demographic and background information such as age, height, history of pain or injury, and descriptions of their physical activity levels. Subjects will receive a clinical screening exam by a licensed physical therapist to determine the type of movement abnormalities present, the severity of their symptoms and to screen for inclusion and exclusion criteria.

To collect scapular position measurement reliability data, subjects will stand through out data collection. Measurements of the scapula will be taken with the mobile application for the arm at rest and in two elevated position. Subjects will wear an off-the-shelf elbow brace when asked to hold their arm in the two elevated positions. These elevated positions will be maintained by having subjects maintain contact of their forearm against a guide. For intra-rater reliability, position measurements will be repeated twice for each of three planes of elevation. Additionally, for inter-rater reliability each measurement will be repeated once by two other examiners. This process will repeated twice when using the application with and without the handle.

For the validation portion of the study, a subgroup of subjects will have the same position measurements performed by a single examiner with additional motion sensors taped to the skin of their scapula and breast bone and a sensor attached to an arm brace strapped to their arm.

In total, the subject will be asked to raise and hold their arm for approximately 5 sec, 36 times during the testing within ranges of motion typically performed during daily activities.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic subjects: subjects without complaints or history of shoulder pain or obvious movement abnormalities.
2. Symptomatic subjects: subjects with shoulder pain who have active range of motion beyond 120° of elevation.

Exclusion Criteria:

1. Symptomatic and asymptomatic subjects: history of trauma including fractures, dislocations, previous shoulder surgeries within the past 6 weeks. Humeral elevation less than 120 degrees, shoulder symptomology that is judged by the examiner to be of cervical origin.
2. Asymptomatic subjects: Complaints of shoulder pain, positive results on joint tests commonly associated with shoulder impingement, presence of shoulder joint movement abnormalities as determined by a physical therapist, including thoracic scoliosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Asymptomatic subjects: subjects without complaints or history of shoulder pain or obvious movement abnormalities.
  2. Symptomatic subjects: subjects with shoulder pain who have active range of motion beyond 120° of elevation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Scapular Position as assessed in degrees of joint angle by the mobile application | baseline
  Scapular position is measured in degrees of joint angle collected by the mobile application software collecting this information from the mobile device's measurement sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Ludewig, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided